CLINICAL TRIAL: NCT00956865
Title: Community Glaucoma Screenings: Assessment of Interventions to Improve Follow-up
Brief Title: Community Glaucoma Screening Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Marlene Moster, MD, Attending Surgeon, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 433
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; Intervention; Follow up
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voucher (Active Comparator): Voucher for transportation reimbursement
  Interventions: Other: Voucher
- Voucher and call (Active Comparator): Voucher for transportation and telephone calls
  Interventions: Other: Voucher; Other: Telephone Call
- Voucher and call and contact (Active Comparator): Voucher for transportation, telephone calls, and a contact at the senior center
  Interventions: Other: Voucher; Other: Telephone Call; Other: Contact

INTERVENTIONS:
Other: Voucher — Vouchers given to reimburse transportation
Other: Telephone Call — Telephone reminder calls
  Arms: Voucher and call; Voucher and call and contact
Other: Contact — Contact at senior center to encourage follow up
  Arms: Voucher and call and contact

SUMMARY:
The purpose of this study is to determine if one of three interventions improves follow-up rates for screening exam participants who are instructed to have a definitive eye exam.

DETAILED DESCRIPTION:
To determine if one of three interventions: vouchers, telephone calls, and personal contacts, improves follow-up rates for screening exam participants who are instructed to have a definitive eye exam.

ELIGIBILITY:
Inclusion Criteria:

* All who had an eye screening exam.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Definitive follow-up eye exam | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Henderer, MD, Principal Investigator — Temple University

IPD SHARING:
Plan to Share IPD: Undecided